CLINICAL TRIAL: NCT03856021
Title: Comparing Outcomes of Microfracture Versus Microfracture and Bone Marrow Aspirate Concentrate for the Treatment of Osteochondral Lesions of the Talus
Brief Title: Microfracture vs. Microfracture and BMAC for Osteochondral Lesions of the Talus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RI2019Shakked
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Osteochondral Lesion of Talus
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microfracture (Active Comparator)
  Interventions: Procedure: Microfracture
- Microfracture with Bone Marrow Aspirate Concentrate (Active Comparator)
  Interventions: Procedure: Microfracture with Bone Marrow Aspirate Concentrate

INTERVENTIONS:
Procedure: Microfracture with Bone Marrow Aspirate Concentrate — Bone Marrow Aspirate Concentrate harvested and prepared from the iliac crest
  Arms: Microfracture with Bone Marrow Aspirate Concentrate
Procedure: Microfracture — All surgeons will use a 2 mm microfracture pick to perform the microfracture procedure. Using the 2 mm pick, surgeons will make 5 holes per 10 cm2.
  Arms: Microfracture

SUMMARY:
Osteochondral lesions of the talus are thought to be due in large part to traumatic events or repetitive microtrauma that causes damage to both the articular cartilage and the subchondral bone. There are several treatment modalities for osteochondral lesions of the talus but there is no consensus as to which is the superior method for repair.

Treatment modalities are aimed at regenerating articular cartilage. Microfracture is a widely accepted and utilized treatment for osteochondral lesions. This procedure results in pluripotent bone marrow stem cells filling the defect and ultimately differentiating into fibrocartilage-producing cells [1]. This technique has shown good results in both short- and medium-term follow-up for smaller lesions. Bone marrow aspirate contains mesenchymal stem cells and growth factors with cartilage regeneration potential. Bone marrow aspirate concentrate (BMAC) is a treatment modality that has shown to have to potential to produce hyaline cartilage. This study aims to analyze the effect of adding BMAC to the standard microfracture procedure in terms of clinical and radiographic outcomes in comparison to patients who only underwent microfracture treatment.

ELIGIBILITY:
Inclusion Criteria:

Greater than 18 years of age and scheduled for surgery to treat osteochondral lesion of the talus Able and willing to sign informed consent document

Exclusion Criteria:

Unwilling to sign informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | 3 years following surgery
  validated patient-reported outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No